CLINICAL TRIAL: NCT01839435
Title: PROSPECTIVE EVALUATION OF OUTPATIENT APPENDECTOMY FOR NON COMPLICATED ACUTE APPENDICITIS: Intention-to-treat Study
Brief Title: Feasibility of Outpatient Appendectomy for Acute Appendicitis
Acronym: APPENDAMBU
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2012_843_0031; 2013-A00170-45 (Other: ID-RCB); 120202B-42 (Other: french ANSM)
Record Dates: First submitted 2013-04-22; First posted 2013-04-24 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Acute Appendicitis
Keywords: appendectomy; acute appendicitis; outpatient
MeSH Terms: conditions — Appendicitis | interventions — Ambulatory Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- outpatient patients (Experimental): Outpatient surgery will be proposed to all patients
  Interventions: Procedure: outpatient surgery

INTERVENTIONS:
Procedure: outpatient surgery

SUMMARY:
The aim of our monocentric prospective in intention-to-treat study is to evaluate the feasibility of outpatient appendectomy for non complicated acute appendicitis.

DETAILED DESCRIPTION:
Acute appendicitis is one of the most common surgical emergencies and corresponds to an high number of admissions (about 120.000) in France. It mainly affects young adults and is associated to fewer complications and to a short length of stay. The notion of outpatient refers to a shorter hospital length to stay i.e. less than 12 hours without an overnight hospitalization. This notion came from 3 learned society recommendations' (SFCD, ACHBT, and AFCA) and has been considered as a national priority.

There is no consensus about appendectomy in an outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* Non complicated acute appendicitis which has been diagnosed at physical, paraclinical and morphological examination
* Adult patient
* Patient with sufficient understanding
* Good compliance with medical prescription
* Hygiene and housing equivalent to a hospitalization
* Availability of an accompanying able to prevent the surgeon if necessary, to accompany the patient and stay at night next to him
* Less than one hour from an health care adapted to the surgical structure
* Quick access to a telephone
* Patient affiliated with social protection

Exclusion Criteria:

* complicated appendicitis
* pregnancy or breastfeeding
* unstable vital signs or fever
* objective signs of diffuse peritonitis
* ward of court or prisoners
* Discovery of a complicated shape (severe sepsis, abscess, generalized peritonitis)
* Discovery of an alternative diagnosis
* Performing an associated gesture (colectomy or typhlectomy, annexectomy...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-04; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
success of outpatient appendectomy | postoperative day 30
  The primary endpoint corresponds to the proportion of outpatient appendectomy defined as the number of patients whose hospital length of stay is less than 12 hours.
  This endpoint will be evaluated during the consult 30 day after the surgery

SECONDARY OUTCOMES:
The unplanned overnight admission rate | postoperative day 30
  the proportion of patients who are discharged more than 12 hours after the surgery and are thus hospitalized for at least one night
The unexpected consultation rate | postoperative day 30
  The unexpected consultation rate reflects the number of AS patients attending the emergency department for a postoperative problem.
The hospital readmission rate | postoperative day 30
  The hospital readmission rate is defined as the number of patients who are discharged from hospital after outpatient surgery but are subsequently readmitted
the reoperation rate | postoperative day 30
  the reoperation rate reflects the proportion of patients who are operated on after their post-outpatient surgery discharge
The proportion of deprogramming | postoperative day 30
  The proportion of deprogramming defined as the number of reconvened patients who do not return the next day
post-surgical pain | the day of the surgery prior to the discharge
  the post-surgical pain is evaluated thanks to the Brief Pain Inventory Form
post-surgical quality of life | the day of the surgery prior to the discharge
  the post-surgical quality of life is evaluated thanks to the SF36 Form

CONTACTS AND LOCATIONS:
Overall Officials: jean marc regimbeau, MD, PhD, Principal Investigator — CHU amiens
Locations (1):
- Amiens University Hospital, Amiens, France

REFERENCES:
- [Background] Sabbagh C, Brehant O, Dupont H, Browet F, Pequignot A, Regimbeau JM. The feasibility of short-stay laparoscopic appendectomy for acute appendicitis: a prospective cohort study. Surg Endosc. 2012 Sep;26(9):2630-8. doi: 10.1007/s00464-012-2244-1. Epub 2012 Mar 23. PMID 22441976
- [Result] Sabbagh C, Masseline L, Grelpois G, Ntouba A, Dembinski J, Regimbeau JM. Management of Uncomplicated Acute Appendicitis as Day Case Surgery: Can Outcomes of a Prospective Study Be Reproduced in Real Life? J Am Coll Surg. 2019 Sep;229(3):277-285. doi: 10.1016/j.jamcollsurg.2019.04.031. Epub 2019 May 13. PMID 31096041